CLINICAL TRIAL: NCT04006119
Title: A Phase II Study of Ad-RTS-hIL-12 + Veledimex in Combination With Cemiplimab-rwlc (Libtayo®) in Subjects With Recurrent or Progressive Glioblastoma
Brief Title: Study of Ad-RTS-hIL-12 + Veledimex in Combination With Cemiplimab in Subjects With Recurrent or Progressive Glioblastoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: Alaunos Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ATI001-204
Record Dates: First submitted 2019-06-28; First posted 2019-07-02 (Actual); Results first posted 2025-04-18 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-03

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — veledimex; cemiplimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ad-RTS-hIL-12 + veledimex in combination with cemiplimab-rwlc (Experimental): Intratumoral Ad-RTS-hIL-12 and oral veledimex (activator ligand, 20mg) given in combination with cemiplimab-rwlc via infusion.
  Interventions: Biological: Ad-RTS-hIL-12; Drug: Veledimex; Drug: Cemiplimab-Rwlc

INTERVENTIONS:
Biological: Ad-RTS-hIL-12 — * intratumoral injection of Ad-RTS-hIL-12
  * 2.0 x 10^11 viral particles (vp) per injection
Drug: Veledimex — 20mg/day 15 oral daily doses of veledimex
Drug: Cemiplimab-Rwlc — Infusion every 3 weeks (350mg)
  Other Names: Libtayo; REGN2810

SUMMARY:
This research study involves an investigational product: Ad-RTS-hIL-12 given with veledimex for production of human IL-12. IL-12 is a protein that can improve the body's natural response to disease by enhancing the ability of the immune system to kill tumor cells and may interfere with blood flow to the tumor.

Cemiplimab-rwlc (Libtayo) is an antibody (a kind of human protein) that is being tested to see if it will allow the body's immune system to work against glioblastoma tumors. Libtayo (cemiplimab-rwlc) is currently FDA approved in the United States for metastatic cutaneous cell carcinoma (CSCC), but is not approved in glioblastoma. Cemiplimab-rwlc may help your immune system detect and attack cancer cells. Ad-RTS-hIL-12 and veledimex will be given in combination with cemiplimab-rwlc to enhance the IL-12 mediated effect observed to date.

The main purpose of this study is to evaluate the safety and efficacy of a single tumoral injection of Ad-RTS-hIL-12 given with oral veledimex in combination with cemiplimab-rwlc.

DETAILED DESCRIPTION:
Eligible patients will receive one dose of cemiplimab-rwlc, via infusion, one week prior to standard of care craniotomy and tumor resection (subtotal or total). On the day of surgery, patients will receive one dose of veledimex before the resection procedure. Ad-RTS-hIL-12 will be administered by free-hand injection. Patients will continue on oral veledimex for 14 days. Following veledimex, patients will receive cemiplimab-rwlc via infusion every three weeks.

The study is divided into three periods: the screening period, the treatment period and the follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject ≥18 and ≤75 years of age
* Provision of written informed consent for tumor resection (subtotal allowed), tumor biopsy, samples collection, and treatment with investigational products prior to undergoing any study-specific procedures
* Histologically confirmed glioblastoma from archival tissue
* Evidence of tumor recurrence/progression by magnetic resonance imaging (MRI) according to Response Assessment in Neuro-Oncology (RANO) criteria after standard initial therapy. Multifocal disease is allowed.
* Previous standard-of-care antitumor treatment including surgery and/or biopsy and chemoradiation. At the time of registration, subjects must have recovered from the toxic effects of previous treatments as determined by the treating physician. The washout periods from prior therapies are intended as follows: (windows other than what is listed below should be allowed only after consultation with the Medical Monitor)

  1. Nitrosoureas: 6 weeks
  2. Other cytotoxic agents: 4 weeks
  3. Antiangiogenic agents: 4 weeks
  4. Targeted agents, including small molecule tyrosine kinase inhibitors: 2 weeks
  5. Vaccine-based or CAR-T therapy: 3 months
* Able to undergo standard MRI scans with contrast agent before enrollment and after treatment
* Karnofsky Performance Status ≥70
* Adequate bone marrow reserves and liver and kidney function, as assessed by the following laboratory requirements:

  1. Hemoglobin ≥9 g/L
  2. Lymphocytes >500/mm3
  3. Absolute neutrophil count ≥1500/mm3
  4. Platelets ≥100,000/mm3
  5. Serum creatinine ≤1.5 x upper limit of normal (ULN)
  6. Aspartate transaminase (AST) and alanine transaminase (ALT) ≤2.5 x ULN
  7. Total bilirubin <1.5 x ULN
  8. International normalized ratio (INR) and activated partial thromboplastin time (aPTT) or partial thromboplastin time (PTT) within normal institutional limits
* Female of child bearing potential* and sexually active male subjects must agree to practice highly effective contraception prior to the start of the first treatment, during the study, and for at least 4 months after the last dose. Highly effective contraceptive measures include stable use of combined (estrogen and progestogen containing) hormonal contraception (oral, intravaginal, transdermal) or progestogen-only hormonal contraception (oral, injectable, implantable) associated with inhibition of ovulation initiated 2 or more menstrual cycles prior to screening; intrauterine device (IUD); intrauterine hormone-releasing system (IUS); bilateral tubal ligation; vasectomized partner; and or sexual abstinence**.

  * Postmenopausal women must be amenorrhoeic for at least 12 months in order not to be considered of childbearing potential. Pregnancy testing and contraception are not required for women with documented hysterectomy or tubal ligation.

  ** Sexual abstinence is considered a highly effective method only if defined as refraining from heterosexual intercourse during the entire period of risk associated with the study treatments. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient.
* Normal cardiac and pulmonary function as evidenced by a normal ECG with QTc ≤450 msec and peripheral oxygen saturation (SpO2) ≥92% on room air by pulse oximetry

Exclusion Criteria:

* Radiotherapy treatment within 4 weeks of starting veledimex
* Prior treatment of disease with bevacizumab (NOTE: short use (< 4 doses) of bevacizumab for controlling edema is allowed)
* Subjects receiving systemic corticosteroids for treatment of disease-related symptoms during the 4 weeks prior to Day -7
* Subjects with clinically significant increased intracranial pressure (e.g., impending herniation or requirement for immediate palliative treatment) or uncontrolled seizures
* Uncontrolled infection with human immunodeficiency virus, hepatitis B or hepatitis C infection; or diagnosis of immunodeficiency. NOTE:

  * Subjects with known HIV infection who have controlled infection (undetectable viral load (HIV RNA PCR) and CD4 count above 350 either spontaneously or on a stable antiviral regimen) are permitted. For Subjects with controlled HIV infection, monitoring will be performed per local standards.
  * Subjects with hepatitis B (HBsAg+) who have controlled infection (serum hepatitis B virus DNA PCR that is below the limit of detection AND receiving anti-viral therapy for hepatitis B) are permitted. Subjects with controlled infections must undergo periodic monitoring of HBV DNA. Patients must remain on anti-viral therapy for at least 6 months beyond the last dose of investigational study drug.
  * Subjects who are hepatitis C virus antibody positive (HCV Ab+) who have controlled infection (undetectable HCV RNA by PCR either spontaneously or in response to a successful prior course of anti-HCV therapy) are permitted.
* Use of systemic antibacterial, antifungal, or antiviral medications for the treatment of acute clinically significant infection within 2 weeks of first veledimex dose. Concomitant therapy for chronic infections is not allowed. Subjects must be afebrile prior to Ad-RTS-hIL-12 injection; only prophylactic antibiotic use is allowed perioperatively.
* Use of enzyme-inducing antiepileptic drugs (EIAED) within 7 days prior to the first dose of study drug. Note: Levetiracetam (Keppra®) is not an EIAED and is allowed.
* Other concurrent clinically active malignant disease, requiring treatment, except for non-melanoma cancers of the skin or carcinoma in situ of the cervix or non-metastatic prostate cancer
* Nursing or pregnant females
* Prior exposure to veledimex
* Use of an investigational product within prior 30 days.
* Prior exposure to inhibitors of immuno-checkpoint pathways (e.g., anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-CTLA-4 antibody) or other agents specifically targeting T cells
* Use of medications that induce, inhibit, or are substrates of CYP450 3A4 prior to veledimex dosing without consultation with the Medical Monitor
* Presence of any contraindication for a neurosurgical procedure
* Use of heparin or other anti-coagulation therapy, or acetylsalicylic acid (ASA), or anti-platelet drug within Day -7 to Day 21 should not be used unless necessary to treat a life-threatening illness. Prophylactic subcutaneous heparin per institutional protocol for prevention of deep vein thrombosis (DVT) may be allowed based on discussion with the Medical Monitor. Concomitant medications should continue to be reviewed in consultation with the Medical Monitor.
* Unstable or clinically significant medical condition that would, in the opinion of the Investigator or Medical Monitor, jeopardize the safety of a subject and/or their compliance with the protocol. Examples include, but are not limited to, a history of myocarditis or congestive heart failure (as defined by New York Heart Association Functional Class III or IV), unstable angina, serious uncontrolled cardiac arrythmia, myocardial infarction within 6 months of screening, active interstitial lung disease (ILD)/pneumonitis or a history of ILD/pneumonitis requiring treatment with systemic steroids uncontrolled asthma, or colitis.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-08-05 (Actual); Study Completion 2021-08-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jaymes Holland, Study Director — Alaunos Therapeutics
Locations (7):
- United States (7):
  - Cedars Sinai, Los Angeles, California
  - University of California - San Francisco, San Francisco, California
  - Baptist MD Anderson Cancer Center, Jacksonville, Florida
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Brigham and Women's, Boston, Massachusetts
  - JFK Medical Center, Edison, New Jersey
  - NYU Langone Health, New York, New York

REFERENCES:
- [Derived] Chiocca EA, Gelb AB, Chen CC, Rao G, Reardon DA, Wen PY, Bi WL, Peruzzi P, Amidei C, Triggs D, Seften L, Park G, Grant J, Truman K, Buck JY, Hadar N, Demars N, Miao J, Estupinan T, Loewy J, Chadha K, Tringali J, Cooper L, Lukas RV. Combined immunotherapy with controlled interleukin-12 gene therapy and immune checkpoint blockade in recurrent glioblastoma: An open-label, multi-institutional phase I trial. Neuro Oncol. 2022 Jun 1;24(6):951-963. doi: 10.1093/neuonc/noab271. PMID 34850166

RESULTS

PARTICIPANT FLOW:
Groups:
- Ad-RTS-hIL-12 + Veledimex in Combination With Cemiplimab-rwlc: Subjects received cemiplimab-rwlc on Day -7 (run in). On Day 0 (day of Ad-RTS-hIL-12 administration) subjects took one dose of veledimex prior to injection of Ad-RTS-hIL-12. After the Ad-RTS-hIL-12 injection, veledimex will be administered orally for 14 days (end of treatment veledimex). Subjects then received a dose of cemiplimab-rwlc on Day 15 and every three weeks thereafter (Q3W) until confirmed progression by immunotherapy Response Assessment for Neuro Oncology (iRANO) criteria (adjuvant cemiplimab) .
Period: Run in Cemiplimab Period
Arm/Group | Ad-RTS-hIL-12 + Veledimex in Combination With Cemiplimab-rwlc
Started | 40
Completed | 39
Not Completed | 1
Not completed — Lack of Efficacy | 1
Period: End of Treatment Veledimex
Arm/Group | Ad-RTS-hIL-12 + Veledimex in Combination With Cemiplimab-rwlc
Started | 39
Completed | 37
Not Completed | 2
Not completed — Adverse Event | 2
Period: Adjuvant Cemiplimab Period
Arm/Group | Ad-RTS-hIL-12 + Veledimex in Combination With Cemiplimab-rwlc
Started | 37
Completed | 0
Not Completed | 37
Not completed — Lack of Efficacy | 28
Not completed — Adverse Event | 3
Not completed — Withdrawal by Subject | 4
Not completed — Sponsor Study Termination rollover to Compassionate Use | 2

BASELINE CHARACTERISTICS:
Population: All subjects who have received at least one dose of any of the investigational agents: cemiplimab-rwlc, Ad-RTS-hIL 12 or veledimex
Groups:
- Ad-RTS-hIL-12 + Veledimex in Combination With Cemiplimab-rwlc: Intratumoral Ad-RTS-hIL-12 and oral veledimex (activator ligand, 20mg) given in combination with cemiplimab-rwlc via infusion.
  Ad-RTS-hIL-12: - intratumoral injection of Ad-RTS-hIL-12
  - 2.0 x 10^11 viral particles (vp) per injection
  Veledimex: 20mg/day 15 oral daily doses of veledimex
  Cemiplimab-Rwlc: Infusion every 3 weeks (350mg)
Arm/Group | Ad-RTS-hIL-12 + Veledimex in Combination With Cemiplimab-rwlc
Number analyzed (Participants) | 40
Age, Continuous [Median (Full Range); unit: Years] | 58 [26 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 25
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 2
  Black or African American | 2
  Caucasian | 35
  Unknown | 1
Region of Enrollment [Number; unit: participants]
  United States | 40
Unifocal Disease [Count of Participants; unit: Participants] | 33
Isocitrate Dehydrogenase wild type (WT) [Count of Participants; unit: Participants] | 37
O6-methlyguanine-DNA methyltransferase (MGMT) unmethylated [Count of Participants; unit: Participants] | 28
Karnofsky performance score (KPS) ≥90 [Count of Participants; unit: Participants] — Patients with better performance status are less likely to experience dose reductions, treatment delays, or early discontinuation, reducing variability in trial outcomes.
  Ethically, trials aim to balance risk and benefit, ensuring that patients are not unduly harmed by enrolling in a study for which they may be too frail and regulatory agencies require trials to include patients who can safely tolerate experimental therapies to ensure valid safety and efficacy assessments.
  Participants | 25

OUTCOME MEASURES:

1. Primary Outcome: Safety of Intratumoral Ad-RTS-hIL-12 and Oral Veledimex in Combination With Cemiplimab-rwlc in Subjects With Recurrent or Progressive Glioblastoma.
Description: Evaluation of adverse events as assessed by CTCAE v5.0 will be based on the incidence, intensity and type of adverse event. Safety evaluations included the observed incidence of treatment-emergent adverse events (TEAEs), serious TEAEs, TEAEs of toxicity Grade >3, TEAEs leading to treatment dose modification, discontinuation, and death. Drug-related TEAEs were also assessed.
Time Frame: 2.0 yrs
Population: The Full Analysis Set (FAS) includes every subject who received at least one dose of any study drug recorded in the Data Management database excluding screen failures.
  The Evaluable Safety Population (ESP) is a subset of the FAS. Regardless of major protocol deviations, these subjects have received at least one of the following:
  * Day -7 of cemiplimab,
  * the injection of Ad-RTS-hIL-12 with at least one post IL-12 dose of veledimex,
  * and at least one post IL-12 dose of cemiplimab (Day 15).
Measure: Number; unit: participants
Arm/Group | Ad-RTS-hIL-12 + Veledimex in Combination With Cemiplimab-rwlc
Number analyzed (Participants) | 40
participants
  Any TEAE | 39
  Any Serious TEAE | 28
  Any TEAE with Toxicity Grade >/= 3 | 32
  Any TEAE Leading to Treatment Discontinuation | 5
  Any TEAE Leading to Death (Progressive Disease) | 8
  Any Drug-Related TEAE | 39
  Any Drug-Related Serious TEAE | 10
  Any Drug-Related TEAE with Toxicity Grade >/=3 | 20
  Any Drug-Related TEAE Leading to Treatment Dose Modification | 11
  Any Drug-Related TEAE Leading to Treatment Discontinuation | 3
  Any Drug-Related TEAE Leading to Death | 0
  Ad-RTS-hIL-12 + Veledimex Related TEAEs | 35
  Ad-RTS-hIL-12 + Veledimex Related Serious TEAEs | 9
  Ad-RTS-hIL-12 + Veledimex Related TEAEs with Toxicity Grade >/= 3 | 17
  Ad-RTS-hIL-12 + Veledimex TEAEs Leading to Treatment Dose Modification | 8
  Ad-RTS-hIL-12 + Veledimex TEAEs Leading to Treatment Discontinuation | 2
  Ad-RTS-hIL-12 + Veledimex Related TEAEs Leading to Death | 0
  Cemiplimab Related TEAEs | 34
  Cemiplimab Related Serious TEAEs | 6
  Cemiplimab Related TEAEs with Toxicity Grade >/= 3 | 17
  Cemiplimab Related TEAEs Leading to Treatment Dose Modification | 3
  Cemiplimab Related TEAEs Leading to Treatment Discontinuation | 1
  Cemiplimab Related TEAEs Leading to Death | 0

2. Primary Outcome: Efficacy of Intratumoral Ad-RTS-hIL-12 and Oral Veledimex in Combination With Cemiplimab-rwlc in Subjects With Recurrent or Progressive Glioblastoma.
Description: Overall Survival (OS)
  OS is defined as the duration of time from the first dose of study drug (i.e., cemiplimab at Day -7) to the date of death from any cause. Censoring will be considered as below:
  * Subjects who discontinue study will be censored at date of discontinuation.
  * Subjects who are lost to follow-up will be censored at last follow-up contact date.
  * If the subject has not died, the subject is censored if still alive up to 2 years from the first dose of study drug received.
Time Frame: 2.0 yrs
Population: The per protocol population will comprise subjects who have received Day -7 of cemiplimab, the injection of Ad-RTS-hIL-12 with at least one post IL-12 dose of veledimex, at least one post IL-12 dose of cemiplimab (e.g. Day 15), and who have not had a major protocol deviation for which the key efficacy endpoints could be regarded as confounded or uninterpretable. Subjects who have had minor protocol deviation(s) that are thought not to impact efficacy will be included in this analysis population.
Measure: Median (Full Range); unit: Months
Arm/Group | Ad-RTS-hIL-12 + Veledimex in Combination With Cemiplimab-rwlc
Number analyzed (Participants) | 37
Months | 12.09 [8.38 to 16.66]

3. Secondary Outcome: To Determine the Survival Rates at 6, 12, and 18 Months
Description: Given the early closure of the study and survival follow-up data limited to one year post last patient in, complete assessment of efficacy could not be determined. Number of participants with death prior to each time point (6, 12, and 18 months) is reported here.
Time Frame: From Day 0 through 18 months post first dose of study treatment
Population: The population will comprise subjects who have received Day -7 of cemiplimab, the injection of Ad-RTS-hIL-12 with at least one post IL-12 dose of veledimex, at least one post IL- 12 dose of cemiplimab (e.g., Day 15), and who have not had a major protocol deviation for which the key efficacy endpoints could be regarded as confounded or uninterpretable. Estimates of the OS at prespecified timepoints will be based on the per protocol (PP) population.
Measure: Number; unit: participants
Arm/Group | Ad-RTS-hIL-12 + Veledimex in Combination With Cemiplimab-rwlc
Number analyzed (Participants) | 37
participants
  Death prior to 6 months | 8
  Death prior to 12 months | 19
  Death prior to 18 months | 24

4. Secondary Outcome: To Determine the Progression Free Survival (PFS)
Description: Given the early closure of the study, formal assessment of PFS using Kaplan Meier Product-Line method was not performed. Mean time to disease progression (or participant's last scan) is reported here.
Time Frame: 2.0 yrs
Population: The per protocol population comprised subjects who had received Day -7 of cemiplimab, the injection of Ad-RTS-hIL-12 with at least 1 post IL-12 dose of veledimex, at least 1 post IL-12 dose of cemiplimab (e.g., Day 15), and who had not had a major protocol deviation for which the key efficacy endpoints could be regarded as confounded or uninterpretable. Subjects who have had minor protocol deviation(s) that are thought not to impact efficacy were included in this analysis population.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Ad-RTS-hIL-12 + Veledimex in Combination With Cemiplimab-rwlc
Number analyzed (Participants) | 39
Days | 89.0 (95.6)

5. Secondary Outcome: To Determine the Rate of Pseudoprogression (PSP) at 6, 12, 18 and 24 Months
Description: Given the early closure of the study complete assessment of efficacy could not be determined. Reported below is the PSP at anytime while on study.
Time Frame: 2 years
Population: Given the early closure of the study complete assessment of efficacy could not be determined. The per protocol population will comprise subjects who have received Day -7 of cemiplimab, the injection of Ad-RTS-hIL-12 with at least one post IL-12 dose of veledimex, at least one post IL-12 dose of cemiplimab (e.g., Day 15), and who have not had a major protocol deviation for which the key efficacy endpoints could be regarded as confounded or uninterpretable.
Measure: Count of Participants; unit: Participants
Arm/Group | Ad-RTS-hIL-12 + Veledimex in Combination With Cemiplimab-rwlc
Number analyzed (Participants) | 37
Participants | 5

6. Secondary Outcome: To Determine the Investigator's Assessment of Response, Including Tumor Objective Response Rate (ORR) at 6, 12, 18 and 24 Months
Description: Tumor response will be defined by radiographic and clinical criteria. Complete response (CR) or partial response (PR) will be first assessed by radiographic changes that indicate a reduction of bi-dimensional tumor size as per Recist 1.1 criteria. In addition, changes in neurologic function and steroid use will be considered to determine stable disease (SD).Given the early closure of the study complete assessment of efficacy could not be determined. The results below report response at anytime while on study.
Time Frame: 2 years
Population: The per protocol population will comprise subjects who have received Day -7 of cemiplimab, the injection of Ad-RTS-hIL-12 with at least one post IL-12 dose of veledimex, at least one post IL-12 dose of cemiplimab (e.g., Day 15), and who have not had a major protocol deviation for which the key efficacy endpoints could be regarded as confounded or uninterpretable.
Measure: Count of Participants; unit: Participants
Arm/Group | Ad-RTS-hIL-12 + Veledimex in Combination With Cemiplimab-rwlc
Number analyzed (Participants) | 37
Participants | 3

7. Secondary Outcome: To Determine the Tumor Response Rates at 6, 12, 18 and 24 Months
Description: Given the early closure of the study and survival follow-up data limited to one year post last patient in, complete assessment of efficacy could not be determined. The IRANO results below report response at anytime while on study.
Time Frame: 2 years
Population: Given the early closure of the study and survival follow-up data limited to one year post last patient in, complete assessment of efficacy could not be determined.
Measure: Count of Participants; unit: Participants
Arm/Group | Ad-RTS-hIL-12 + Veledimex in Combination With Cemiplimab-rwlc
Number analyzed (Participants) | 37
Participants | 3

8. Secondary Outcome: Changes From Baseline in Cellular Responses Elicited by Ad-RTS-hIL-12 and Veledimex in Combination With Cemiplimab-rwlc
Description: Immune cell population markers, such as cluster of differentiation (CD) antigens CD3+CD4+ and CD3+/ CD4+/ CD25hi/ Foxp3+/ CD127lo-, were assessed.
Time Frame: Screening through Day 28 (assessed at Screening and Days 0, 1, 3, 7, 14, and 28)
Population: The biomarker-evaluable population includes all ESP subjects who have adequate biomarker sample(s) at screening (baseline) and at least one follow-up assessment
Measure: Mean (Standard Deviation); unit: % of total lymphocytes
Arm/Group | Ad-RTS-hIL-12 + Veledimex in Combination With Cemiplimab-rwlc
Number analyzed (Participants) | 29
% of total lymphocytes
  CD3+CD4+ at Screening: number analyzed (Participants) | 24
  CD3+CD4+ at Screening | 40.85 (10.42)
  CD3+CD4+ at Day 0: number analyzed (Participants) | 26
  CD3+CD4+ at Day 0 | 40.26 (11.28)
  CD3+CD4+ at Day 1: number analyzed (Participants) | 17
  CD3+CD4+ at Day 1 | 35.36 (12.38)
  CD3+CD4+ at Day 3: number analyzed (Participants) | 19
  CD3+CD4+ at Day 3 | 46.85 (12.38)
  CD3+CD4+ at Day 7: number analyzed (Participants) | 22
  CD3+CD4+ at Day 7 | 39.96 (7.81)
  CD3+CD4+ at Day 14: number analyzed (Participants) | 21
  CD3+CD4+ at Day 14 | 33.00 (12.28)
  CD3+CD4+ at Day 28: number analyzed (Participants) | 17
  CD3+CD4+ at Day 28 | 37.17 (11.54)
  CD3+/ CD4+/ CD25hi/ Foxp3+/ CD127lo- at Screening: number analyzed (Participants) | 24
  CD3+/ CD4+/ CD25hi/ Foxp3+/ CD127lo- at Screening | 0.67 (0.60)
  CD3+/ CD4+/ CD25hi/ Foxp3+/ CD127lo- at Day 0: number analyzed (Participants) | 26
  CD3+/ CD4+/ CD25hi/ Foxp3+/ CD127lo- at Day 0 | 0.82 (0.64)
  CD3+/ CD4+/ CD25hi/ Foxp3+/ CD127lo- at Day 1: number analyzed (Participants) | 17
  CD3+/ CD4+/ CD25hi/ Foxp3+/ CD127lo- at Day 1 | 0.44 (0.46)
  CD3+/ CD4+/ CD25hi/ Foxp3+/ CD127lo- at Day 3: number analyzed (Participants) | 19
  CD3+/ CD4+/ CD25hi/ Foxp3+/ CD127lo- at Day 3 | 1.02 (0.81)
  CD3+/ CD4+/ CD25hi/ Foxp3+/ CD127lo- at Day 7: number analyzed (Participants) | 22
  CD3+/ CD4+/ CD25hi/ Foxp3+/ CD127lo- at Day 7 | 0.55 (0.51)
  CD3+/ CD4+/ CD25hi/ Foxp3+/ CD127lo- at Day 14: number analyzed (Participants) | 21
  CD3+/ CD4+/ CD25hi/ Foxp3+/ CD127lo- at Day 14 | 0.50 (0.49)
  CD3+/ CD4+/ CD25hi/ Foxp3+/ CD127lo- at Day 28: number analyzed (Participants) | 17
  CD3+/ CD4+/ CD25hi/ Foxp3+/ CD127lo- at Day 28 | 0.48 (0.47)

9. Secondary Outcome: Changes From Baseline in Humoral Immune Responses Elicited by Ad-RTS-hIL-12 and Veledimex in Combination With Cemiplimab-rwlc
Description: Immunological and biological markers, such as levels of interleukin-12 (IL-12) and interferon gamma (IFN-γ) were assessed in serum samples.
Time Frame: Screening through Day 28 (assessed at Screening and Days 0, 1, 3, 7, 14, and 28)
Population: The biomarker-evaluable population includes all Evaluable Safety Population (ESP) subjects who have adequate biomarker sample(s) at screening (baseline) and at least one follow-up assessment. Individual samples that were below the limit of quantitation were considered 0.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Ad-RTS-hIL-12 + Veledimex in Combination With Cemiplimab-rwlc
Number analyzed (Participants) | 27
pg/mL
  IFN-gamma at Screening | 0.00 (0.00)
  IFN-gamma at Day 0: number analyzed (Participants) | 26
  IFN-gamma at Day 0 | 0.11 (0.58)
  IFN-gamma at Day 1: number analyzed (Participants) | 22
  IFN-gamma at Day 1 | 0.18 (0.83)
  IFN-gamma at Day 3: number analyzed (Participants) | 24
  IFN-gamma at Day 3 | 10.53 (20.34)
  IFN-gamma at Day 7: number analyzed (Participants) | 21
  IFN-gamma at Day 7 | 6.43 (13.12)
  IFN-gamma at Day 14: number analyzed (Participants) | 21
  IFN-gamma at Day 14 | 0.74 (2.04)
  IFN-gamma at Day 28: number analyzed (Participants) | 19
  IFN-gamma at Day 28 | 10.07 (42.86)
  IL-12 at Screening | 0.00 (0.00)
  IL-12 at Day 0: number analyzed (Participants) | 26
  IL-12 at Day 0 | 0.09 (0.48)
  IL-12 at Day 1: number analyzed (Participants) | 22
  IL-12 at Day 1 | 0.28 (0.73)
  IL-12 at Day 3: number analyzed (Participants) | 24
  IL-12 at Day 3 | 29.65 (49.96)
  IL-12 at Day 7: number analyzed (Participants) | 21
  IL-12 at Day 7 | 15.56 (23.09)
  IL-12 at Day 14: number analyzed (Participants) | 21
  IL-12 at Day 14 | 6.80 (12.24)
  IL-12 at Day 28: number analyzed (Participants) | 19
  IL-12 at Day 28 | 31.06 (131.49)

ADVERSE EVENTS:
Time Frame: 2 year
Groups:
- Ad-RTS-hIL-12 + Veledimex in Combination With Cemiplimab-rwlc: Ad-RTS-hIL-12 and oral veledimex (activator ligand, 20 mg) given in combination with cemiplimab-rwlc via infusion. One dose of cemiplimab-rwlc on Day -7, then every 3 weeks starting on Day 15
Arm/Group | Ad-RTS-hIL-12 + Veledimex in Combination With Cemiplimab-rwlc
All-Cause Mortality (participants affected / at risk) | 24/40
Serious Adverse Events (participants affected / at risk) | 30/40
Other Adverse Events (participants affected / at risk) | 39/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ad-RTS-hIL-12 + Veledimex in Combination With Cemiplimab-rwlc (N=40)
Aphasia (Nervous system disorders) | 2 (2)
Brain abscess (Infections and infestations) | 1 (1)
Brain oedema (Nervous system disorders) | 4 (4)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1)
COVID-19 (Infections and infestations) | 2 (2)
Cytokine release syndrome (Immune system disorders) | 1 (1)
Disease progression (General disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Embolism (Vascular disorders) | 1 (1)
Encephalopathy (Nervous system disorders) | 5 (5)
Enterocolitis (Gastrointestinal disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (3)
Female genital tract fistula (Reproductive system and breast disorders) | 1 (1)
Gait disturbance (General disorders) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 2 (2)
Headache (Nervous system disorders) | 4 (4)
Hemiparesis (Nervous system disorders) | 2 (2)
Hydrocephalus (Nervous system disorders) | 2 (2)
Hypernatraemia (Metabolism and nutrition disorders) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 1 (1)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5)
Meningitis (Infections and infestations) | 1 (1)
Mental disorder (Psychiatric disorders) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1)
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Neutrophil count decreased (Investigations) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1)
Postoperative wound infection (Infections and infestations) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pyrexia (General disorders) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1)
Seizure (Nervous system disorders) | 4 (4)
Sepsis (Infections and infestations) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1)
Wound infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ad-RTS-hIL-12 + Veledimex in Combination With Cemiplimab-rwlc (N=40)
Abdominal pain (Gastrointestinal disorders) | 3 (3)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Abulia (Psychiatric disorders) | 1 (1)
Acidosis (Metabolism and nutrition disorders) | 1 (1)
Acquired diaphragmatic eventration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Action tremor (Nervous system disorders) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 1 (2)
Agitation (Psychiatric disorders) | 3 (5)
Alanine aminotransferase increased (Investigations) | 8 (13)
Amylase increased (Investigations) | 2 (3)
Anaemia (Blood and lymphatic system disorders) | 8 (10)
Androgen deficiency (Endocrine disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 3 (3)
Aphasia (Nervous system disorders) | 18 (27)
Apraxia (Nervous system disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (6)
Aspartate aminotransferase increased (Investigations) | 8 (9)
Asthenia (General disorders) | 2 (3)
Ataxia (Nervous system disorders) | 2 (2)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Atrial flutter (Cardiac disorders) | 1 (1)
Autonomic nervous system imbalance (Nervous system disorders) | 1 (1)
Bacteraemia (Infections and infestations) | 1 (1)
Balance disorder (Nervous system disorders) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 1 (1)
Blood bilirubin increased (Investigations) | 2 (2)
Blood calcium decreased (Investigations) | 2 (2)
Blood glucose increased (Investigations) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 7 (8)
Blood magnesium decreased (Investigations) | 1 (1)
Blood phosphorus decreased (Investigations) | 1 (1)
Blood potassium decreased (Investigations) | 3 (4)
Blood pressure increased (Investigations) | 1 (2)
Blood sodium decreased (Investigations) | 2 (3)
Blood sodium increased (Investigations) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1)
Brain oedema (Nervous system disorders) | 1 (1)
Carpal tunnel syndrome (Nervous system disorders) | 1 (1)
Chills (General disorders) | 3 (3)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Clumsiness (Nervous system disorders) | 1 (1)
Cognitive disorder (Nervous system disorders) | 4 (5)
Confusional state (Psychiatric disorders) | 8 (10)
Constipation (Gastrointestinal disorders) | 16 (18)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
C-reactive protein increased (Investigations) | 5 (6)
Cystitis (Infections and infestations) | 1 (1)
Cytokine release syndrome (Immune system disorders) | 2 (4)
Decreased appetite (Metabolism and nutrition disorders) | 4 (4)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Delirium (Psychiatric disorders) | 2 (2)
Depression (Psychiatric disorders) | 2 (2)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 2 (2)
Device related thrombosis (General disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 8 (9)
Disturbance in attention (Nervous system disorders) | 2 (2)
Dizziness (Nervous system disorders) | 7 (7)
Dry eye (Eye disorders) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (3)
Dysarthria (Nervous system disorders) | 3 (4)
Dysgeusia (Nervous system disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 4 (4)
Dysphagia (Gastrointestinal disorders) | 4 (6)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Ear discomfort (Ear and labyrinth disorders) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (1)
Ear pruritus (Ear and labyrinth disorders) | 1 (1)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Encephalopathy (Nervous system disorders) | 5 (5)
Erythema (Skin and subcutaneous tissue disorders) | 1 (2)
Facial paralysis (Nervous system disorders) | 3 (3)
Facial paresis (Nervous system disorders) | 4 (4)
Fall (Injury, poisoning and procedural complications) | 7 (13)
Fatigue (General disorders) | 14 (16)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 3 (3)
Gait disturbance (General disorders) | 3 (4)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Gaze palsy (Eye disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 2 (4)
Haemorrhage intracranial (Nervous system disorders) | 3 (4)
Haemorrhoids (Gastrointestinal disorders) | 1 (1)
Hallucination (Psychiatric disorders) | 1 (1)
Headache (Nervous system disorders) | 23 (40)
Hemianopia (Nervous system disorders) | 1 (1)
Hemianopia homonymous (Nervous system disorders) | 2 (2)
Hemiparesis (Nervous system disorders) | 11 (18)
Hordeolum (Infections and infestations) | 1 (2)
Hydrocephalus (Nervous system disorders) | 1 (1)
Hyperamylasaemia (Metabolism and nutrition disorders) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 10 (21)
Hypersomnia (Nervous system disorders) | 1 (1)
Hypertension (Vascular disorders) | 9 (10)
Hyperthyroidism (Endocrine disorders) | 5 (5)
Hypoaesthesia (Nervous system disorders) | 2 (2)
Hypocalcaemia (Metabolism and nutrition disorders) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 10 (15)
Hyponatraemia (Metabolism and nutrition disorders) | 11 (15)
Hypophagia (Metabolism and nutrition disorders) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 8 (8)
Hypotension (Vascular disorders) | 5 (6)
Hypothyroidism (Endocrine disorders) | 9 (9)
Incision site discharge (Injury, poisoning and procedural complications) | 1 (1)
Incision site pain (Injury, poisoning and procedural complications) | 2 (2)
Influenza (Infections and infestations) | 1 (1)
Influenza like illness (General disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 7 (7)
International normalised ratio increased (Investigations) | 2 (2)
Irritability (Psychiatric disorders) | 2 (4)
Lactic acidosis (Metabolism and nutrition disorders) | 1 (1)
Lethargy (Nervous system disorders) | 4 (5)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Lipase (Investigations) | 1 (1)
Lipase increased (Investigations) | 3 (3)
Localised oedema (General disorders) | 2 (2)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lymphocyte count decreased (Investigations) | 15 (41)
Lymphopenia (Blood and lymphatic system disorders) | 6 (11)
Malaise (General disorders) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 1 (1)
Memory impairment (Nervous system disorders) | 5 (5)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1)
Mobility decreased (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Mutism (Psychiatric disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 23 (34)
Nervous system disorder (Nervous system disorders) | 1 (1)
Neuralgia (Nervous system disorders) | 2 (3)
Neurologic neglect syndrome (Nervous system disorders) | 1 (1)
Neutrophil count decreased (Investigations) | 4 (5)
Nocturia (Renal and urinary disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Occipital neuralgia (Nervous system disorders) | 1 (1)
Oedema peripheral (General disorders) | 4 (4)
Onychomycosis (Infections and infestations) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Otitis externa (Infections and infestations) | 1 (1)
Pain (General disorders) | 2 (2)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1)
Paraesthesia (Nervous system disorders) | 4 (7)
Penile pain (Reproductive system and breast disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Peroneal nerve palsy (Nervous system disorders) | 1 (1)
Personality change (Psychiatric disorders) | 1 (1)
Platelet count decreased (Investigations) | 5 (9)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumocephalus (Injury, poisoning and procedural complications) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 2 (2)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1)
Procedural headache (Injury, poisoning and procedural complications) | 7 (7)
Procedural pain (Injury, poisoning and procedural complications) | 5 (6)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3)
Pseudomeningocele (Injury, poisoning and procedural complications) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pyrexia (General disorders) | 25 (40)
Rash (Skin and subcutaneous tissue disorders) | 2 (3)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 6 (7)
Red blood cell sedimentation rate increased (Investigations) | 3 (3)
Respiratory rate increased (Investigations) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Secondary adrenocortical insufficiency (Endocrine disorders) | 1 (1)
Seizure (Nervous system disorders) | 7 (7)
Sensory loss (Nervous system disorders) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 3 (4)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 (2)
Skin laceration (Injury, poisoning and procedural complications) | 2 (2)
Somnolence (Nervous system disorders) | 2 (3)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 4 (4)
Temperature intolerance (General disorders) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 2 (2)
Tongue geographic (Gastrointestinal disorders) | 1 (1)
Transaminases increased (Investigations) | 1 (1)
Tremor (Nervous system disorders) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 3 (3)
Urinary retention (Renal and urinary disorders) | 6 (8)
Urinary tract infection (Infections and infestations) | 6 (9)
Visual field defect (Nervous system disorders) | 5 (6)
Vomiting (Gastrointestinal disorders) | 14 (15)
Weight decreased (Investigations) | 6 (6)
Weight decreased (Investigations) | 8 (10)
White blood cell count increased (Investigations) | 1 (1)
Wound infection (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2020-01-08): https://cdn.clinicaltrials.gov/large-docs/19/NCT04006119/Prot_000.pdf
  • Statistical Analysis Plan (2021-08-18): https://cdn.clinicaltrials.gov/large-docs/19/NCT04006119/SAP_001.pdf